CLINICAL TRIAL: NCT02455440
Title: Esmolol Reduces Anesthetic Requirements Thereby Facilitating Early Extubation; a Prospective Controlled Study in Patients Undergoing Intracranial Surgery
Brief Title: Esmolol Infusion in Patients Undergoing Craniotomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: George Papanicolaou Hospital (Other)
Responsible Party: Principal Investigator, Asouhidou Irene, Dr.Irene Asouhidou, George Papanicolaou Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GeorgePH
Record Dates: First submitted 2015-05-09; First posted 2015-05-27 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Cerebral Arterial Disease; Cerebral Aneurysm
Keywords: esmolol; anesthetics
MeSH Terms: conditions — Cerebral Arterial Diseases; Intracranial Aneurysm | interventions — esmolol; Propofol; Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Esmolol (Active Comparator): 500 mcg/kg of esmolol bolus 10 min before induction of anesthesia, followed by additional 200 mcg/kg/min of esmolol until 30 minutes after extubation.
  Interventions: Drug: Esmolol; Drug: Propofol and sevoflurane
- control (Placebo Comparator): Control group did not receive esmolol or other b-blocker in the perioperative period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esmolol — effect of esmolol on intraoperative fluctuations of propofol and sevoflurane. Propofol and sevoflurane intraoperative concentration will be expressed as mean ± SD. Differences in categorical data will be evaluated using the student t test.
  Other Names: propofol; sevoflurane
  Arms: Esmolol
Drug: Placebo
  Arms: control
Drug: Propofol and sevoflurane
  Arms: Esmolol

SUMMARY:
Anesthesia techniques that minimize anesthetic requirements and their effects may be beneficial. Esmolol, a short acting hyperselective β-adrenergic blocker is effective in blunting adrenergic response to several perioperative stimuli and so it might interfere in the effect of the anesthetic drugs on the brain. This study was designed to investigate the effect of esmolol on the consumption of propofol and sevoflurane in patients undergoing craniotomy.

DETAILED DESCRIPTION:
Patients undergoing elective craniotomy for aneurysm clipping or tumor dissection were randomly divided in two groups (four subgroups). Anesthesia was induced with propofol, fentanyl and a single dose of cis-atracurium, followed by continuous infusion of remifentanil and either propofol or sevoflurane. Patients in the esmolol group received 500 mcg/kg of esmolol bolus 10 min before induction of anesthesia, followed by additional 200 mcg/kg/min of esmolol. Monitoring of the depth of anesthesia was also performed using the Bispectral Index-BIS. It was also performed monitoring of the cardiac output in order to evaluate the effect of esmolol on cardiac output.

The inspired concentration of sevoflurane and the infusion rate of propofol were adjusted in order to maintain a BIS value between 40-50.

Intraoperative emergence was detected by the elevation of BIS value, HR or MAP.

It was recorded intraoperative fluctuations of propofol and sevoflurane in both groups. Data were expressed as mean ± SD. Differences in categorical data were evaluated using the student t test.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA physical status 1-3
* Glasgow Coma Scale:15

Exclusion Criteria:

* Patients with ASA physical status >3,
* Body Mass Index (BMI) over 30,
* indication for rapid sequence induction,
* any contraindication for receiving b-blocker,
* chronic use of b-blocker,
* Glasgow Coma Scale (GCS) <15,
* history of drug abuse,
* severe mental impairment,
* preoperative aphasia,
* neurologic deficit or preoperatively foreseen delayed extubation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
systolic arterial pressure fluctuation | intraoperative

SECONDARY OUTCOMES:
extubation time | at time of surgery
Heart rate | intraoperative
effect of esmolol on anesthetic's concentration | intraoperative

CONTACTS AND LOCATIONS:
Locations (1):
- George Papanikolaou General Hospital, Thessaloniki, Thessaloniki, Greece

REFERENCES:
- [Background] Wilson ES, McKinlay S, Crawford JM, Robb HM. The influence of esmolol on the dose of propofol required for induction of anaesthesia. Anaesthesia. 2004 Feb;59(2):122-6. doi: 10.1111/j.1365-2044.2004.03460.x. PMID 14725513
- [Background] Grillo P, Bruder N, Auquier P, Pellissier D, Gouin F. Esmolol blunts the cerebral blood flow velocity increase during emergence from anesthesia in neurosurgical patients. Anesth Analg. 2003 Apr;96(4):1145-1149. doi: 10.1213/01.ANE.0000055647.54957.77. PMID 12651674
- [Background] Bilotta F, Lam AM, Doronzio A, Cuzzone V, Delfini R, Rosa G. Esmolol blunts postoperative hemodynamic changes after propofol-remifentanil total intravenous fast-track neuroanesthesia for intracranial surgery. J Clin Anesth. 2008 Sep;20(6):426-30. doi: 10.1016/j.jclinane.2008.04.006. PMID 18929282
- [Derived] Asouhidou I, Trikoupi A. Esmolol reduces anesthetic requirements thereby facilitating early extubation; a prospective controlled study in patients undergoing intracranial surgery. BMC Anesthesiol. 2015 Nov 28;15:172. doi: 10.1186/s12871-015-0154-1. PMID 26615516